CLINICAL TRIAL: NCT05598762
Title: The Transcriptomic Study of Thai Patients With Atopic Dermatitis by Tape Strips
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queen Sirikit National Institute of Child Health (Other Government)
Collaborators: Mahidol University (Other); Icahn School of Medicine at Mount Sinai (Other); Samitivej Hospital group (Unknown)
Responsible Party: Principal Investigator, Tassalapa Daengsuwan, Assistant Professor, Queen Sirikit National Institute of Child Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 65-007
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Atopic Dermatitis
Keywords: tape strips; endotype
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Children with mild atopic dermatitis (Active Comparator): * age 1-8 years old
  * mild degree of atopic dermatitis
  Interventions: Genetic: Tape strips
- Children with moderate-severe atopic dermatitis (Active Comparator): * age 1-8 years old
  * moderate or severe degree of atopic dermatitis
  Interventions: Genetic: Tape strips
- Children with food allergy and moderate-severe atopic dermatitis (Active Comparator): * age 1-8 years old
  * moderate or severe degree of atopic dermatitis
  * IgE mediated food allergy
  Interventions: Genetic: Tape strips
- Adult with atopic dermatitis (Active Comparator): * age 18-60 years old
  * mild-severe atopic dermatitis
  Interventions: Genetic: Tape strips
- Healthy (Active Comparator): * age 1-60 years old
  * no history of atopic diseases
  Interventions: Genetic: Tape strips
- Healthy with Asthma (Active Comparator): * age 1-8 years old
  * doctor diagnosed asthma
  * no history of chronic or chronic relapsing eczema
  Interventions: Genetic: Tape strips

INTERVENTIONS:
Genetic: Tape strips — Tape strip is a minimally invasive method that captures the stratum corneum. It is use to identify skin biomarkers in atopic dermatitis.

SUMMARY:
This study will be use the tape strip technique to evaluate the skin biomarkers of atopic dermatitis among Thai patients to differentiate clinical phenotype.

DETAILED DESCRIPTION:
The patients will be enrolled in this study if they have been diagnosed with atopic dermatitis. All participants (AD patients and controls) will be evaluated their skin biomarkers by using tape stripping. The tape strips will be applied to the antecubital fossa to collect the epithelial samples. Then RNA was extracted from the tape strips for mRNA profiling to identify the immune and epidermal barrier genes.

ELIGIBILITY:
Inclusion Criteria:

* Children (age 1-18 years old) with mild atopic dermatitis
* Children (age 1-18 years old) with moderate to severe atopic dermatitis
* Children (age 1-18 years old) with moderate to severe atopic dermatitis and food allergy
* Adult (age 18-60 years old) with atopic dermatitis
* Healthy individuals (1-60 years old)
* Patients with asthma (1-60 years old)

Exclusion Criteria:

* Active skin infections
* Used systemic immunosuppressants within 4 weeks
* Used topical steroids or immunomodulators within 1 week
* Used moisturizers within 12 hours before evaluation

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Cellular AD biomarkers | 1 month
  Evaluated by RNA sequencing: RNA was extracted for real-time polymerase chain reaction (RT-PCR) with the miRNAeasy Mini Kit (Qiagen, Hilden, Germany). Reverse transcription to complementary DNA (cDNA) from RNA was carried out using the High Capacity cDNA reverse transcription (Thermo fisher). TaqMan Low Density Array (TLDA) cards (Thermo fisher) were used for quantitative reverse transcription polymerase chain reaction (qRT-PCR). 500pg total RNA was used for PreAMP pool. Eukaryotic 18S recombinant RNA (rRNA) was used as an endogenous control. Expression values were normalized to Rplp0
Immune biomarkers | 1 month
  Evaluated by RNA sequencing: RNA was extracted for real-time polymerase chain reaction (RT-PCR) with the miRNAeasy Mini Kit (Qiagen, Hilden, Germany). Reverse transcription to complementary DNA (cDNA) from RNA was carried out using the High Capacity cDNA reverse transcription (Thermo fisher). TaqMan Low Density Array (TLDA) cards (Thermo fisher) were used for quantitative reverse transcription polymerase chain reaction (qRT-PCR). 500pg total RNA was used for PreAMP pool. Eukaryotic 18S recombinant RNA (rRNA) was used as an endogenous control. Expression values were normalized to Rplp0
Barrier biomarkers | 1 month
  chain reaction (RT-PCR) with the miRNAeasy Mini Kit (Qiagen, Hilden, Germany). Reverse transcription to complementary DNA (cDNA) from RNA was carried out using the High Capacity cDNA reverse transcription (Thermo fisher). TaqMan Low Density Array (TLDA) cards (Thermo fisher) were used for quantitative reverse transcription polymerase chain reaction (qRT-PCR). 500pg total RNA was used for PreAMP pool. Eukaryotic 18S recombinant RNA (rRNA) was used as an endogenous control. Expression values were normalized to Rplp0

CONTACTS AND LOCATIONS:
Overall Officials: Panipak Temboonnark, MD, Principal Investigator — Queen Sirikit National Institute of Child Health
Locations (1):
- Queen Sirikit National Institute of Child Health, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Czarnowicki T, He H, Krueger JG, Guttman-Yassky E. Atopic dermatitis endotypes and implications for targeted therapeutics. J Allergy Clin Immunol. 2019 Jan;143(1):1-11. doi: 10.1016/j.jaci.2018.10.032. PMID 30612663
- [Result] Brunner PM, Guttman-Yassky E. Racial differences in atopic dermatitis. Ann Allergy Asthma Immunol. 2019 May;122(5):449-455. doi: 10.1016/j.anai.2018.11.015. Epub 2018 Nov 20. PMID 30465859
- [Result] Chan TC, Sanyal RD, Pavel AB, Glickman J, Zheng X, Xu H, Cho YT, Tsai TF, Wen HC, Peng X, Cueto I, Krueger JG, Guttman-Yassky E. Atopic dermatitis in Chinese patients shows TH2/TH17 skewing with psoriasiform features. J Allergy Clin Immunol. 2018 Sep;142(3):1013-1017. doi: 10.1016/j.jaci.2018.06.016. Epub 2018 Jun 28. No abstract available. PMID 29964056
- [Result] Guttman-Yassky E, Diaz A, Pavel AB, Fernandes M, Lefferdink R, Erickson T, Canter T, Rangel S, Peng X, Li R, Estrada Y, Xu H, Krueger JG, Paller AS. Use of Tape Strips to Detect Immune and Barrier Abnormalities in the Skin of Children With Early-Onset Atopic Dermatitis. JAMA Dermatol. 2019 Dec 1;155(12):1358-1370. doi: 10.1001/jamadermatol.2019.2983. PMID 31596431